CLINICAL TRIAL: NCT06343974
Title: Noninvasive Evaluation of Fetal Hyperinsulinemia With Ultrasound Radiomics
Status: Recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Mikael Huhtala, Physician, MD, PhD, Turku University Hospital
Other Study IDs: 0843
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy in Diabetic; Diabetes Mellitus, Type 1
Keywords: ultrasonography; fetus; radiomics; hyperinsulinemia; liver; pregnancy
MeSH Terms: conditions — Pregnancy in Diabetics; Diabetes Mellitus, Type 1; Hyperinsulinism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 diabetes: Pregnant woman with type 1 diabetes.
- Healthy controls: Pregnant women with uncomplicated pregnancy and normal oral glucose tolerance test (OGTT).

SUMMARY:
The goal of this observational study is to compare fetal liver ultrasound radiomics between pregnancies complicated by type 1 diabetes and healthy controls.

The main questions it aims to answer are:

* Are fetal liver ultrasound radiomic features reproducible?
* Does fetal liver ultrasound radiomics differ between pregnancies complicated by type 1 diabetes and healthy controls?

Participants will undergo ultrasound examination to collect ultrasound data for the analyses.

DETAILED DESCRIPTION:
Gestational diabetes is a growing health concern posing the neonate in the risk of adverse outcomes, such as macrosomia, cesarean delivery, hypoglycemia, respiratory morbidity, and need for neonatal intensive care. Most of these outcomes are either closely or causally related to fetal hyperinsulinemia, which is induced by maternal hyperglycemia. However, the accurate and non-invasive means of estimating fetal hyperinsulinemia are currently lacking.

Given that maternal diabetes and fetal hyperinsulinemia are associated with profound changes in fetal liver blood supply, biometry, metabolism, and lipid content, it was hypothesized that fetal hyperinsulinemia would be detectable by ultrasound using modern computer-aided technologies, i.e., radiomics and machine learning. In this prospective pilot study, the aim is to recruit 20 pregnant women with type I diabetes and compare them to 40 healthy controls. Patients with type 1 diabetes were chosen because their pregnancies are known to be associated with fetal hyperinsulinemia. Study subjects will be recruited at Turku University Hospital and the City of Turku maternity welfare clinics. It is assumed that radiomics analysis of fetal liver ultrasound pictures will indicate fetal hyperinsulinemia in pregnancies complicated by type 1 diabetes at 34 gestational weeks. Simultaneously, the inter- and intraobserver variability for fetal liver ultrasound radiomic features will be characterized.

In the future, non-invasive evaluation of fetal hyperinsulinemia could provide a useful tool in managing pregnancies complicated by maternal diabetes - either pre-gestational or gestational.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years
* Capable to give an informed consent
* Singleton pregnancy
* Planning to deliver in Turku University Hospital
* Maternal BMI < 40
* Gestational age should be confirmed by first trimester ultrasound
* Normal oral glucose tolerance test (OGTT) at 24-28 gestational weeks in controls

Exclusion Criteria:

* Major fetal chromosomal, genetic, or structural anomaly
* Fetal growth restriction, or birth weight < 10th centile
* Birth weight > 90th centile or polyhydramnios in the controls
* Non-reassuring fetal status requiring immediate treatment, or intrauterine fetal demise
* Verified fetal infection (e.g. cytomegalovirus, toxoplasma, hepatitis B and C), excluding bacterial infection due to intrapartum chorioamnionitis
* Placenta accreta spectrum disorder
* Major maternal medical condition requiring systemic pharmacological treatment, other than non-severe hypertension, hypothyroidism, asthma, mild psychiatric disorders, etc.
* Alcohol or tobacco use, or substance abuse in pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women will be recruited at Turku University Hospital and Turku maternity welfare clinics during their routine pregnancy follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Fetal liver ultrasound texture | 34+0 - 34+6 weeks of gestation
  Fetal liver ultrasound texture is the collection of radiomic features that are extracted from the fetal liver ultrasound picture. The ultrasound pictures are acquired using transabdominal ultrasound. The radiomic features are extracted using conventional radiomics libraries e.g. pyradiomics.

SECONDARY OUTCOMES:
Birth weight in grams | After delivery, up to 24 hours
  Birth weight in grams as routinely measured after birth.
Birth weight centile | After delivery, up to 24 hours
  Birth weight adjusted for gestational age, fetal sex, and maternal parity.
Large for gestational age (LGA) | After delivery, up to 24 hours
  Birth weight above 90th centile
Interventricular septum (IVS) width | 34+0 - 34+6 weeks of gestation
  Fetal cardiac interventricular septum (IVS) width, measured at 34 gestational weeks
Number of pregnancies with neonatal hypoglycemia | During initial hospitalization, up to one week of age
  Neonatal plasma glucose < 2.6 mmol/L
Rate of neonatal hypoglycemia treated with oral dextrose gel | During initial hospitalization, up to three weeks of age
  Neonatal plasma glucose < 2.6 mmol/L and treatment with oral dextrose gel
Rate of neonatal hypoglycemia treated with intravenous (IV) glucose | During initial hospitalization, up to three weeks of age
  Neonatal plasma glucose < 2.6 mmol/L and treatment with IV glucose
Length of treatment for neonatal hypoglycemia | During initial hospitalization, up to three weeks of age
  Length of dextrose gel or IV glucose treatment (days)
Number of neonates admitted to neonatal intensive care unit (NICU) | During initial hospitalization, up to one week of age
  Neonatal admission to NICU
Length of NICU admission | During initial hospitalization, up to the age of three months
  Length of NICU admission (days)
Number of pregnancies with neonatal respiratory complications related to maternal diabetes | During initial hospitalization, up to one week of age
  Diagnosis of respiratory distress syndrome and/or transient tachypnea of the newborn
Number of pregnancies with neonatal hyperbilirubinemia | During initial hospitalization, up to two weeks of age
  Neonatal hyperbilirubinemia requiring phototherapy
Maternal HbA1c concentration | Close to 12, 21 and 32 weeks of gestation
  Maternal HbA1c (mmol/mol)
Glucose management indicator (GMI) | Close to 12, 21 and 32 weeks of gestation
  HbA1c estimation based on continuous glucose monitoring (CGM) or flash glucose monitoring data
Time in glycemic range (TIR) | Close to 12, 21 and 32 weeks of gestation
  Time in glycemic range (TIR), if using CGM or flash monitoring
Time above glucose range | Close to 12, 21 and 32 weeks of gestation
  Time above glucose range, if using CGM or flash monitoring
Time below glucose range | Close to 12, 21 and 32 weeks of gestation
  Time below glucose range, if using CGM or flash monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Huhtala, M.D., Ph.D., Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
To ensure study subject anonymity the study data will not be published.